CLINICAL TRIAL: NCT00622050
Title: The Effects of Limiting TV Viewing on Diet, Exercise, and Sleep in Overweight and Obese Adults
Brief Title: The Relationship of TV Viewing to Energy Balance in Adults
Acronym: TView
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Jean Harvey-Berino/ Chair, Department of Nutrition and Food Sciences, Universtiy of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHRBS 08-052
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental): This arm will be experiencing the same protocol as the control group, only their TV viewing time will be reduced. The TV viewing time reduction is the experimental intervention.
  Interventions: Behavioral: TV viewing reduction
- Control (Active Comparator): The control group will be experiencing the exact protocol; only their TV viewing time will not be reduced.
  Interventions: Behavioral: No TV viewing reduction

INTERVENTIONS:
Behavioral: No TV viewing reduction — In the control group, no intervention will be acted upon. This group will receive the exact same protocol as the intervention group, but with observation only.
  Arms: Control
Behavioral: TV viewing reduction — In the experimental arm, TV viewing time will be reduced for half of the study protocol time (3-4 weeks of a 6-8 week protocol).
  Arms: 1

SUMMARY:
The specific objectives of this project are to:

1. Investigate the effects of reducing TV viewing time on energy intake, eating behavior, and energy expenditure in overweight or obese adult subjects, thus providing a basis for evaluating if reducing TV viewing time might be a useful adjunct therapy in obesity prevention and treatment
2. Analyze the types of foods eaten in conjunction with TV viewing
3. Determine if there is an association between location of TV and BMI.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25-50
* Watch at least 3 hours of TV per day or 21 hours per week.
* Between the ages of 21-65 years.
* Willing to have study staff enter home several times.
* Willing to have TV viewing time reduced.

Exclusion Criteria:

* Live greater than 45 minutes from UVM campus.
* Enrolled in a weight loss study
* Pregnant or planning to become pregnant during active study protocol.
* Breastfeeding for 6 months or less.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Energy Intake | Phase I and Phase II

SECONDARY OUTCOMES:
Energy expenditure | Phase I and Phase II

CONTACTS AND LOCATIONS:
Locations (1):
- UVM Department of Nutrition and Food Sciences, Burlington, Vermont, United States

REFERENCES:
- [Derived] Otten JJ, Jones KE, Littenberg B, Harvey-Berino J. Effects of television viewing reduction on energy intake and expenditure in overweight and obese adults: a randomized controlled trial. Arch Intern Med. 2009 Dec 14;169(22):2109-15. doi: 10.1001/archinternmed.2009.430. PMID 20008695
- [Derived] Otten JJ, Littenberg B, Harvey-Berino JR. Relationship between self-report and an objective measure of television-viewing time in adults. Obesity (Silver Spring). 2010 Jun;18(6):1273-5. doi: 10.1038/oby.2009.371. Epub 2009 Oct 29. PMID 19875989
- See also: Website for interested subjects — http://uvm.edu/~tview